CLINICAL TRIAL: NCT04803214
Title: ReActiv8 Stimulation Therapy vs Optimal Medical Management: A Randomized Evaluation
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mainstay Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 980012
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain
Keywords: Neurostimulation; Stimulation; Multifidus; Restorative neurostimulation; Multifidus muscle control; Neurostimulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (ReActiv8) (Active Comparator): Market-approved ReActiv8 device
  Interventions: Device: ReActiv8
- Control (OMM) (No Intervention): Optimized medical management (OMM) (Standard of Care)

INTERVENTIONS:
Device: ReActiv8 — Market-approved ReActiv8 device implanted
  Arms: Treatment (ReActiv8)

SUMMARY:
This study is a prospective, randomized study comparing ReActiv8 Therapy to Optimal Medical Management (OMM).

DETAILED DESCRIPTION:
This study is a prospective, randomized study comparing ReActiv8 Therapy to Optimal Medical Management (OMM), where OMM means the patient is managed according to available guideline-directed treatments (e.g., medication, physical therapy, injections) individualized to meet the patient needs. All patients who satisfy the enrollment criteria are randomized (1:1) to receive either ReActiv8 (Treatment group) or OMM (Control group).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years
2. Evidence of lumbar multifidus muscle dysfunction
3. Intractable Chronic Low Back Pain that has persisted >6 months resulting in pain most of the days in the past 12 months
4. Failed therapy including pain medications and physical therapy
5. Not a candidate for spine surgery
6. Low Back Pain NRS of ≥6 and ≤9
7. Oswestry Disability Index score ≥30 and ≤60
8. Willing and capable of giving Informed Consent
9. Able to comply with this protocol
10. On Optimal Medical Management per the Investigator

Exclusion Criteria:

1. Contraindicated for the ReActiv8 System
2. BMI > 35
3. Any surgical correction procedure for scoliosis at any time, or a current clinical diagnosis of moderate to severe scoliosis
4. An independent MRI assessment identifying a pathology that is likely the cause of the CLBP and is amenable to surgery
5. Leg pain described as being worse than back pain, or radiculopathy (neuropathic pain) below the knee
6. Any condition unrelated to CLBP which, in the opinion of the Investigator, could limit physical movement or compliance with the protocol, or interfere with the assessment of efficacy
7. Surgical and other procedure exclusions
8. Psycho-social exclusions
9. Protocol compliance exclusions
10. General exclusions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2026-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Schwab, Study Chair — New York-Presbyterian; Chris Gilligan, Study Chair — Brigham and Women's Hospital; Kiran Patel, Study Chair — Northwell Health
Locations (28):
- United States (28):
  - Barrow Brain & Spine, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - SoCal Sport and Spine, Newport Beach, California
  - Pacific Research Institute, Santa Rosa, California
  - University of Colorado, Aurora, Colorado
  - International Spine, Pain and Performance Center, Washington D.C., District of Columbia
  - Cleveland Clinic Martin Health Tradition Hospital, Port Saint Lucie, Florida
  - Cantor Spine Center and Paley Orthopedic Spine Institute, West Palm Beach, Florida
  - Augusta Orthopedic & Sports Medicine Specialists, Augusta, Georgia
  - Horizon Clinical Research, Fayetteville, Georgia
  - Vista Clinical Research, Newnan, Georgia
  - Indiana Spine Group, Carmel, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Advent Health Shawnee Mission, Shawnee Mission, Kansas
  - Columbia Orthopedic Group, Columbia, Missouri
  - SSM Health Medical Group, Jefferson City, Missouri
  - Freeman Hospital, Joplin, Missouri
  - Northwell Health, Great Neck, New York
  - Ainsworth Institute of Pain Management, New York, New York
  - OrthoCarolina Sports Medicine Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Pacific Sports and Spine, Eugene, Oregon
  - Spinal Diagnostics, PC, Tualatin, Oregon
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilligan C, Burnside D, Grant L, Yong RJ, Mullins PM, Schwab F, Mekhail N. ReActiv8 Stimulation Therapy vs. Optimal Medical Management: A Randomized Controlled Trial for the Treatment of Intractable Mechanical Chronic Low Back Pain (RESTORE Trial Protocol). Pain Ther. 2023 Apr;12(2):607-620. doi: 10.1007/s40122-023-00475-4. Epub 2023 Feb 14. PMID 36787013
- [Result] Schwab F, Mekhail N, Patel KV, Langhorst M, Heros RD, Gentile J, Costandi S, Moore G, Gilmore C, Manion S, Chakravarthy K, Meyer SC, Bundy JV, Tate JL, Sanders R, Vaid S, Szentirmai O, Goree J, Patel VV, Lehmen J, Desai MJ, Pope JE, Giuffrida A, Hayek S, Virk SS, Paicius R, Klemme WR, Levy R, Gilligan C; RESTORE investigators. Restorative Neurostimulation Therapy Compared to Optimal Medical Management: A Randomized Evaluation (RESTORE) for the Treatment of Chronic Mechanical Low Back Pain due to Multifidus Dysfunction. Pain Ther. 2025 Feb;14(1):401-423. doi: 10.1007/s40122-024-00689-0. Epub 2025 Jan 15. PMID 39812968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 386 participants were screened across 25 clinical sites. The first participant was enrolled in July 2021 and the last participant was enrolled in July 2023.
Pre-assignment Details: Of the 386 participants screened, 203 were randomized and attended at least one follow-up visit. The protocol and analysis plan required randomized patients attend at least one follow-up visit to be included in analyses.
Groups:
- Treatment (ReActiv8): Participants were treated with restorative neurostimulation (ReActiv8) which consists of two 30-minute stimulation sessions per day at the L2 medial branch of the dorsal ramus in addition to continued OMM through 1 year
  Stimulation frequency: 20 Hz
- Control (OMM): A treatment plan consisting of non-investigational interventions (e.g., pharmacological agents, physical or psychosocial therapies) individualized to each patient's specific needs that was established prior to randomization through 1 year. Optimal medical management (OMM).
Period: Overall Study
Arm/Group | Treatment (ReActiv8) | Control (OMM)
Started | 99 | 104
1.5 Month Follow up | 97 (2 patients missed visit) | 99 (5 patients missed visit)
3 Month Follow up | 96 (3 patients missed visit) | 97 (6 patients missed visit)
6 Month Follow up | 95 (3 patients missed visit) | 98 (4 patients missed visit)
12 Month Follow up | 94 | 94 (3 patients missed visit)
Completed | 94 | 94
Not Completed | 5 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Missed 12 month visit | 0 | 3

BASELINE CHARACTERISTICS:
Population: Number of subjects who were randomized and attended at least one follow-up visit
Groups:
- Control (OMM): A treatment plan consisting of non-investigational interventions (e.g., pharmacological agents, physical or psychosocial therapies) individualized to each patient's specific needs that was established prior to randomization through 1 year
- Total: Total of all reporting groups
Arm/Group | Treatment (ReActiv8) | Control (OMM) | Total
Number analyzed (Participants) | 99 | 104 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11) | 48 (13) | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 68 | 126
  Male | 41 | 36 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — U.S. National Institutes of Health (NIH) and U.S. Office of Management and Budget (OMB) Classification Categories
  Participants
    Hispanic or Latino | 4 | 4 | 8
    Not Hispanic or Latino | 95 | 100 | 195
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — U.S. National Institutes of Health (NIH) and U.S. Office of Management and Budget (OMB) Classification Categories
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 92 | 97 | 189
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 99 | 104 | 203
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29 (4) | 28 (4) | 29 (4)
Pain duration (years from first occurrence) [Mean (Standard Deviation); unit: years] | 11.8 (9.7) | 11.1 (7.5) | 11.4 (8.7)
Percent of Days with low back pain (LBP) in the last 12 months [Mean (Standard Deviation); unit: % of days] | 95 (13) | 97 (8) | 96 (11)
Leg pain [Count of Participants; unit: Participants] | 31 | 28 | 59
LBP NRS [Mean (Standard Deviation); unit: units on a scale] — Low back pain (LBP) numeric rating scale (NRS) is measured on a scale of 0 to 10 where a lower score is a better outcome.
  units on a scale | 7.1 (0.8) | 7.1 (0.9) | 7.1 (0.9)
EQ-5D-5L index score [Mean (Standard Deviation); unit: units on a scale] — European Quality of Life 5-Dimensions 5 Level (EQ-5D-5L) is measured on a scale of -0.5 to 1.0 where a higher score is a better outcome.
  units on a scale | 0.626 (0.116) | 0.612 (0.125) | 0.619 (0.120)
ODI [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index (ODI) is measured on a scale of 0 to 100 where a lower score is a better outcome.
  units on a scale | 44 (8) | 44 (8) | 44 (8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Oswestry Disability Index (ODI)
Description: Comparison of 1-year change from baseline in ODI between Treatment and Control with MMRM for missing data.
  ODI is measured on a scale of 0 to 100 where a lower score is a better outcome.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (ReActiv8) | Control (OMM)
Number analyzed (Participants) | 99 | 104
units on a scale | -19.7 (1.4) | -2.9 (1.4)
Statistical Analysis 1: Comparison: Treatment (ReActiv8) vs Control (OMM); Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Low Back Pain Numerical Rating Scale (LBP NRS)
Description: Comparison of 1-year change from baseline in LBP NRS between Treatment and Control with MMRM for missing data.
  NRS is measured on a scale of 0 to 10 where a higher score is a better outcome.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (ReActiv8) | Control (OMM)
Number analyzed (Participants) | 99 | 104
score on a scale | -3.6 (0.2) | -0.6 (0.2)
Statistical Analysis 1: Comparison: Treatment (ReActiv8) vs Control (OMM); Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change in EQ-5D
Description: Comparison of 1-year change from baseline in EQ-5D between Treatment and Control with MMRM for missing data.
  EQ-5D is measured on a scale of -0.5 to 1.0 where a higher score is a better outcome.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (ReActiv8) | Control (OMM)
Number analyzed (Participants) | 99 | 104
score on a scale | 0.155 (0.012) | 0.008 (0.012)
Statistical Analysis 1: Comparison: Treatment (ReActiv8) vs Control (OMM); Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (ReActiv8) | Control (OMM)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/104
Serious Adverse Events (participants affected / at risk) | 7/99 | 1/104
Other Adverse Events (participants affected / at risk) | 22/99 | 10/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ReActiv8) (N=99) | Control (OMM) (N=104)
Pocket infection (Infections and infestations) | 1 (1) | 0 (0) — Implant site pocket infection
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Aneurysm cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aseptic Meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhagic stroke (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Eye disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ReActiv8) (N=99) | Control (OMM) (N=104)
Device overstimulation of tissue (Product Issues) | 5 (5) | 0 (0)
Implant site pocket pain (Surgical and medical procedures) | 8 (9) | 0 (0)
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (11)

LIMITATIONS AND CAVEATS:
Participants were not blinded to their treatment, and as a result, those randomized to the control arm may have experienced a nocebo effect underestimating the clinical effect of OMM. In addition, patients in the treatment arm may have experienced a placebo effect after being randomized to interventional treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04803214/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04803214/SAP_001.pdf